CLINICAL TRIAL: NCT03074487
Title: Exploratory Study Regarding the Use of Neurophysiological Monitoring Techniques to Detect Spinal Cord Ischemia in Patients After Thoracoabdominal Aortic Aneurysm Repair
Brief Title: Evaluating Monitoring Techniques for Postoperative Spinal Cord Ischemia
Acronym: SINATRA
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL58137.068.16
Record Dates: First submitted 2017-02-21; First posted 2017-03-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Monitoring; Postoperative; Spinal Cord Ischemia; Thoracoabdominal Aneurysm; TAAA; NIRS; Long Loop Reflexes; F-waves
Keywords: Spinal cord ischemia; Postoperative; Thoracoabdominal Aneurysm; Monitoring
MeSH Terms: conditions — Spinal Cord Ischemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Near-infrared spectroscopy
  Other Names: NIRS
Device: Long loop reflex measurements
  Other Names: F-waves

SUMMARY:
During open surgery of a thoraco-abdominal aortic aneurysma (TAAA), diminished blood flow to the myelum can result in hypoxia, compromising proper function of the spinal cord.

Intraoperatively, motor evoked potentials (MEP) are elicited to measure the functional integrity of the spinal cord. MEPs have proven to be a reliable marker of spinal cord ischemia. Moreover, these potentials react within minutes, which facilitates interventions to restore the blood flow. Monitoring intraoperatively with this ancillary test has reduced the rate of paraparesis to < 5%. Unfortunately, in the early postoperative period, spinal cord vulnerability is high. Therefore, some patients develop paraparesis, not during the surgical procedure, but after the surgical procedure. Postoperatively, suboptimal blood flow may lead to critical loss of function. This inadequate perfusion results in "delayed paraparesis". In the postoperative patient, it is not possible to measure MEPs when sedation is decreased, due to the high intensity of the electrical stimulus, which is unacceptably painful in the unanesthetized or partially anesthetized patient. Therefore ancillary tests are needed which can detect spinal cord ischemia postoperatively early, thus preceding the phase with clinically overt paraparesis. The test should be reliable and easy to perform for an extended period of time (up to several days).

The purpose of this study is to explore the usefulness of various neurophysiological tests regarding accuracy and feasibility for the detection of spinal cord ischemia. In particular, to find a diagnostic test which is acceptable for the unanesthetized or partially anesthetized patient and therefore can also be performed postoperatively. These tests will be examined in fully sedated as well as partially sedated patients.

The following candidate tests will be examined:

1. Long loop reflexes (LLR) consisting of F-waves.
2. Oxygenation measurements of the paraspinal muscles using Near-infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Thoraco-abdominal aneurysm (TAA) of the descending aorta: Crawford type I,II, III, IV or V
* Repair using open surgical or endovascular procedure.
* Undergoing monitoring by motor evoked potentials (MEP) as part of the standard surgical procedure.

Exclusion Criteria:

* Aneurysm only in ascending part of the aorta
* Standard contraindications for motor evoked potential (MEP) monitoring.
* Standard contraindications for electrode placement (skin wounds, etc.)
* No informed consent can be obtained prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a thoraco-abdominal aortic aneurysm (TAAA) repair by either open surgical or endovascular procedures are eligible for inclusion. The study population will include patients undergoing TAAA repair in Maastricht (Netherlands), Aachen (Germany) and Bern, (Switzerland).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2025-04 (Actual)

PRIMARY OUTCOMES:
changes in MEP signals perioperative | 8 hours
  These signals will be recoded into categorical variables. To determine associations logistic regression analysis will be performed (univariate and multivariate adjusting for confounders). Screening test calculations (sensitivity, specificity, positive and negative predictive values, false-positive and false-negative rates) will be performed using standard contingency table methods. Agreement between the methods (vs MEP) will be estimated using the Cohen k statistic. The results will first be evaluated descriptively to fine-tune the cut-off values in de the definitive protocol.
Presence of LLR (F-waves) perioperative | 8 hours
  These signals will be recoded into categorical variables. To determine associations logistic regression analysis will be performed (univariate and multivariate adjusting for confounders). Screening test calculations (sensitivity, specificity, positive and negative predictive values, false-positive and false-negative rates) will be performed using standard contingency table methods. Agreement between the methods (vs MEP) will be estimated using the Cohen k statistic. The results will first be evaluated descriptively to fine-tune the cut-off values in de the definitive protocol.
Oxygenation of the paraspinal muscle tissue measured by NIRS perioperative | 8 hours
  These signals will be recoded into categorical variables. To determine associations logistic regression analysis will be performed (univariate and multivariate adjusting for confounders). Screening test calculations (sensitivity, specificity, positive and negative predictive values, false-positive and false-negative rates) will be performed using standard contingency table methods. Agreement between the methods (vs MEP) will be estimated using the Cohen k statistic. The results will first be evaluated descriptively to fine-tune the cut-off values in de the definitive protocol.

SECONDARY OUTCOMES:
The occurrence of intra- and postoperative changes in LLR (F-waves) | 24 hours
  These signals will be recoded into categorical variables. To determine associations logistic regression analysis will be performed (univariate and multivariate adjusting for confounders). Screening test calculations (sensitivity, specificity, positive and negative predictive values, false-positive and false-negative rates) will be performed using standard contingency table methods. The results will first be evaluated descriptively to fine-tune the cut-off values in de the definitive protocol.
The occurrence intra- and postoperative changesNIRS of the paraspinal muscle tissue | 24 hours
  These signals will be recoded into categorical variables. To determine associations logistic regression analysis will be performed (univariate and multivariate adjusting for confounders). Screening test calculations (sensitivity, specificity, positive and negative predictive values, false-positive and false-negative rates) will be performed using standard contingency table methods. The results will first be evaluated descriptively to fine-tune the cut-off values in de the definitive protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacobs MJ, Mess W, Mochtar B, Nijenhuis RJ, Statius van Eps RG, Schurink GW. The value of motor evoked potentials in reducing paraplegia during thoracoabdominal aneurysm repair. J Vasc Surg. 2006 Feb;43(2):239-46. doi: 10.1016/j.jvs.2005.09.042. PMID 16476594
- [Background] Greiner A, Mess WH, Schmidli J, Debus ES, Grommes J, Dick F, Jacobs MJ. Cyber medicine enables remote neuromonitoring during aortic surgery. J Vasc Surg. 2012 May;55(5):1227-32; discussion 1232-3. doi: 10.1016/j.jvs.2011.11.121. Epub 2012 Feb 15. PMID 22341581
- [Background] Armstrong KL, Wood D. Can infant death from child abuse be prevented? Med J Aust. 1992 Feb 17;156(4):290. doi: 10.5694/j.1326-5377.1992.tb139757.x. No abstract available. PMID 1738333
- [Background] Etz CD, Di Luozzo G, Zoli S, Lazala R, Plestis KA, Bodian CA, Griepp RB. Direct spinal cord perfusion pressure monitoring in extensive distal aortic aneurysm repair. Ann Thorac Surg. 2009 Jun;87(6):1764-73; discussion 1773-4. doi: 10.1016/j.athoracsur.2009.02.101. PMID 19463592
- [Background] Jacobs MJ, Mess WH. The role of evoked potential monitoring in operative management of type I and type II thoracoabdominal aortic aneurysms. Semin Thorac Cardiovasc Surg. 2003 Oct;15(4):353-64. doi: 10.1053/s1043-0679(03)00084-4. PMID 14710377
- [Background] Etz CD, von Aspern K, Gudehus S, Luehr M, Girrbach FF, Ender J, Borger M, Mohr FW. Near-infrared spectroscopy monitoring of the collateral network prior to, during, and after thoracoabdominal aortic repair: a pilot study. Eur J Vasc Endovasc Surg. 2013 Dec;46(6):651-6. doi: 10.1016/j.ejvs.2013.08.018. Epub 2013 Sep 5. PMID 24099957
- [Background] Moerman A, Van Herzeele I, Vanpeteghem C, Vermassen F, Francois K, Wouters P. Near-infrared spectroscopy for monitoring spinal cord ischemia during hybrid thoracoabdominal aortic aneurysm repair. J Endovasc Ther. 2011 Feb;18(1):91-5. doi: 10.1583/10-3224.1. PMID 21314355
- [Background] Boezeman RP, van Dongen EP, Morshuis WJ, Sonker U, Boezeman EH, Waanders FG, de Vries JP. Spinal near-infrared spectroscopy measurements during and after thoracoabdominal aortic aneurysm repair: a pilot study. Ann Thorac Surg. 2015 Apr;99(4):1267-74. doi: 10.1016/j.athoracsur.2014.10.032. Epub 2015 Jan 14. PMID 25596871